CLINICAL TRIAL: NCT01164020
Title: Creatine Supplementation and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Creatine and Cognition
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Cognition; Aging
Keywords: cognition; supplementation creatine; resistance training; aging
MeSH Terms: interventions — Creatine; Glucose; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo control (Placebo Comparator): this only receives placebo (dextrose)
  Interventions: Other: Placebo (Dextrose)
- placebo and exercise (Experimental): this is trained and receives placebo
  Interventions: Other: Placebo (Dextrose); Other: Resistance training
- creatine supplementation (Experimental): this is non-exercise trained and receives creatine supplementation
  Interventions: Dietary Supplement: creatine supplementation
- Creatine and Exercise (Experimental): this is exercised trained and receives creatine supplementation
  Interventions: Dietary Supplement: creatine supplementation; Other: Resistance training

INTERVENTIONS:
Dietary Supplement: creatine supplementation — 20g/d for 7 days followed by 5g/d for 23 weeks
  Arms: Creatine and Exercise; creatine supplementation
Other: Placebo (Dextrose) — 20g/d for 7 days followed by 5g/d for 23 weeks
  Arms: placebo and exercise; placebo control
Other: Resistance training — resistance training twice a week for 24 weeks
  Arms: Creatine and Exercise; placebo and exercise

SUMMARY:
Resistance training as well as creatine supplementation may be beneficial for cognitive function, such as memory and attention. Therefore, the investigators speculate that resistance training combined with creatine supplementation would promote additive benefits on cognitive function in elderly women.

ELIGIBILITY:
Inclusion Criteria:

* women older than 60 years old

Exclusion Criteria:

* cardiovascular diseases or muscular disturbances precluding exercise training
* drugs affecting the cognition

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
cognitive function | six months

SECONDARY OUTCOMES:
physical capacity | six months
  muscle strength and function

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Principal Investigator — University of Sao Paulo; Antonio H Lancha Junior, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Medicine - Division of Rheumatology, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Alves CR, Merege Filho CA, Benatti FB, Brucki S, Pereira RM, de Sa Pinto AL, Lima FR, Roschel H, Gualano B. Creatine supplementation associated or not with strength training upon emotional and cognitive measures in older women: a randomized double-blind study. PLoS One. 2013 Oct 3;8(10):e76301. doi: 10.1371/journal.pone.0076301. eCollection 2013. PMID 24098469